CLINICAL TRIAL: NCT00743639
Title: Autologous Transplantation of Bone Marrow Mononuclear Stem-Cells for Dilated Cardiomyopathy: Randomized Clinical Trial
Brief Title: Autologous Transplantation of Bone Marrow Mononuclear Stem-Cells for Dilated Cardiomyopathy
Acronym: SDILCM
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Instituto de Cardiologia do Rio Grande do Sul (Other)
Collaborators: Fundação de Amparo à Pesquisa do Estado do Rio Grande do Sul, Brazil (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: James Fracasso, Instituto de Cardiologia do Rio Grande do Sul / Fund. Universit. Cardiologia
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UP3758
Record Dates: First submitted 2008-08-28; First posted 2008-08-29 (Estimated); Last update posted 2008-08-29 (Estimated); Status verified 2008-06

CONDITIONS: Dilated Cardiomyopathy
Keywords: Cardiomyopathy; stem cell; cardiac failure
MeSH Terms: conditions — Cardiomyopathy, Dilated; Cardiomyopathies; Heart Failure

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Other): Interventional
  Interventions: Procedure: intramyocardial bone marrow stem cells implantation

INTERVENTIONS:
Procedure: intramyocardial bone marrow stem cells implantation — Control group: the patients will be monitored with regular medical visits. Echocardiography: baseline,3,6,9 months. Cardiac NMR at baseline, 3 and 9 months.
  Interventional group: Bone-marrow was collected from in the anterior-superior iliac crest and mononuclear stem cells were isolated by centrifugation in the density rate Ficoll-Hypaque 1.077 media. Technique - The approach was through a left mini-thoracotomy. Twenty small injections of cellular suspension were directly made through a 21F butterfly needle(total=5ml), in the anterior, lateral, posterior and apical faces of the LV ((average 9.6±2.6 x 10[7] cells). After the procedure, the patients were kept in the p.o. for a minimum period of 24hrs. They were released from the hospital in a period that varied from 5-7 days.

SUMMARY:
This study describes a controlled randomized clinical trial to evaluate the efficacy of bone marrow derived stem-cell implants by minithoracotomy in patients with dilated cardiomyopathy and cardiac failure class III or NYHA.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis made at more than one year and symptomatic at functional class III-IV by the New York Heart Association classification (NYHA) despite optimal pharmacologic therapy
* Left ventricular ejection fraction (LVEF) less than 35% by echocardiogram
* Age below 70 years
* Absence of neoplasm
* Abscence of hematologic disease or systemic disease
* No previous cardiac intervention

Exclusion Criteria:

* Episodes of tachycardia or ventricular fibrillation
* Severe or moderated mitral insufficiency
* Any other valvulopathies
* Previous cardiac surgery

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2005-07; Primary Completion 2006-06 (Actual); Study Completion 2008-06 (Actual)

PRIMARY OUTCOMES:
Increase of the ejection function of the left ventricle | twelve months

CONTACTS AND LOCATIONS:
Overall Officials: Renato AK Kalil, MD, PhD, Study Director — Institute of Cardiology of Rio Grande do Sul / FUC
Locations (1):
- Institute of Cardiology of Rio Grande do Sul / FUC, Porto Alegre, Rio Grande do Sul, Brazil